CLINICAL TRIAL: NCT04139772
Title: A Randomized Multicenter Phase III Trial Comparing Docetaxel or Hormone Therapy as Second Line Treatment in Patients With Asymptomatic or Oligosymptomatic Metastatic Castration-resistent Prostate Cancer (mCRPC) Progressing After Abiraterone or Enzalutamide.
Brief Title: Docetaxel or Hormone Therapy as Second Line Treatment in Patients With Asymptomatic or Oligosymptomatic Metastatic Castration-resistent Prostate Cancer (mCRPC) Progressing After Abiraterone or Enzalutamide.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meet-Uro4
Record Dates: First submitted 2019-09-30; First posted 2019-10-25 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Castration-resistent Prostate Cancer
Keywords: metastatic castration-resistent prostate cancer; asymptomatic or oligosymptomatic; hormone therapy; docetaxel
MeSH Terms: interventions — Docetaxel; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Comparative Randomized Phase 3 Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Active Comparator): Docetaxel 75 mg/m2 intravenous (iv) infusion every 3 weeks plus oral prednisone 5 mg twice daily for a maximum of 10 cycles.
  Interventions: Drug: Docetaxel
- Abiraterone or Enzalutamide (Experimental): Patient will receive Abiraterone or Enzalutamide based on previous treatment.
  Abiraterone given orally at the dose of 1000 mg daily plus oral prednisone 5 mg twice daily until progression or unacceptable toxicity. One course of therapy corresponds to four weeks of treatment.
  Enzalutamide given orally at the dose of 160 mg daily until progression or unacceptable toxicity. One course of therapy corresponds to four weeks of treatment.
  Interventions: Drug: Abiraterone Acetate or Enzalutamide

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg/m2 intravenous (iv) infusion every 3 weeks plus oral prednisone 5 mg twice daily for a maximum of 10 cycles.
  Arms: Docetaxel
Drug: Abiraterone Acetate or Enzalutamide — Patient will receive Abiraterone or Enzalutamide based on previous treatment.
  Abiraterone given orally at the dose of 1000 mg daily plus oral prednisone 5 mg twice daily until progression or unacceptable toxicity. One course of therapy corresponds to four weeks of treatment.
  Enzalutamide given orally at the dose of 160 mg daily until progression or unacceptable toxicity. One course of therapy corresponds to four weeks of treatment.
  Arms: Abiraterone or Enzalutamide

SUMMARY:
This is a randomized phase 3 trial aiming to compare the efficacy of docetaxel and hormone therapy as second line treatment in patients with mCRPC progressing after therapy with abiraterone or enzalutamide.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive docetaxel or hormone therapy (abiraterone or enzalutamide based on previous treatment).

Docetaxel (standard) will be administered for 10 cycles (maximum).

Hormone therapy (experimental) will be administered until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Distant metastatic disease
* Previous first line treatment with abiraterone or enzalutamide for 6 cycles interrupted at least 2 weeks before randomization
* Patients must be ≥ 18 years of age
* Patients must have castrate serum level of testosterone of < 0.5 ng/mL ( 1.7 nmol/L)
* Asymptomatic or Oligosymptomatic disease
* Progressive disease according to Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
* ECOG performance status (PS) of 0-2
* Sexually active males must use an accepted and effective method birth control measure
* Written informed consent

Exclusion Criteria:

* Prior exposure to docetaxel or abiraterone for treatment of hormone-sensitive metastatic prostate cancer (mHSPC)
* History of adrenal insufficiency or hypoaldosteronism
* Any medical condition that would make prednisone use contraindicated
* Any medical condition that would make docetaxel use contraindicated
* Patients unable to swallow orally administered medication
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) requiring antiretroviral therapy
* Other malignancy within the last 5 years, except for adequately treated non melanoma skin cancer, bladder cancer (pTis, pTa, pT1) or other solid tumours curatively treated with no evidence of disease for > 5 years
* Participation in another clinical study with an investigational product within 30 days prior to randomization
* Persistent toxicities [>Common Terminology Criteria for Adverse Event (CTCAE) grade 1)] caused by previous cancer therapy prior to randomization
* Uncontrolled medical conditions including diabetes mellitus. Clinically significant cardiovascular disease (e.g.: uncontrolled hypertension or arrhythmia, unstable angina pectoris, congestive heart failure (CHF), vascular disease (arterial thrombosis) and myocardial infarction within < 6 months
* Left ventricular ejection fraction < 50%
* Peripheral neuropathy [> CTCAE grade 2]
* Inadequate bone marrow function defined as:

  * haemoglobin < 9.0 g/dL
  * absolute neutrophils count (ANC) <1.5 x 109/L (> 1500 per mm3)
  * platelet count <100 x 109/L (>100,000 per mm3)
* Inadequate renal and hepatic function, defined as:

  * total serum bilirubin > 1,0 x ULN
  * AST/SGOT o ALT/SGPT > 1,5 x ULN
  * calculated creatinine clearance < 40 mL/min
  * potassium level < 3,5 mmol/L
  * Child-Pugh class C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with metastatic castration resistent prostate cancer
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 5 years
  OS is defined as the time from randomization until death

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 5 years
  PFS is defined as the time elapsed from the date of randomization to the date of progression, as defined by investigators, or the date of death, whichever comes first.
Time to Prostate-Specific Antigen (PSA) Progression | up to 5 years
  as determined by investigator
Incidence of symptomatic skeletal events (SSE) | up to 5 years
  reporting the incidence and types of skeletal related events
Time to symptomatic skeletal event (SSE) | up to 5 years
  Time from the date of randomization to the date of documented symptomatic skeletal event
Time to Pain Progression | up to 5 years
  Time from the date of randomization to the date of pain progression
Number of participants with treatment-related side effects as assessed by Common Terminology Criteria for Adverse Event (CTCAE) version 5.0 | baseline, during treatment (every 4 weeks) up to 5 years
  graded according to Common Terminology Criteria for Adverse Event (CTCAE) version 5.0
Determination of changes in quality of life | baseline, during treatment up to 5 years
  EORTC QLQ-C30, a quality of life questionnaires, composed by 30 items graded from1 (not at all) to 4 (very much) after 1 year from the diagnosis
Radiographic response (bone lesions) | up to 5 years
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Radiographic response (soft tissue lesions) | up to 5 years
  Prostate Cancer Working Group 3 (PCWG3) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD, PhD, Principal Investigator — National Cancer Institute, Naples; Gaetano Facchini, MD, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, MD, PhD, Principal Investigator — National Cancer Institute, Naples; Orazio Caffo, MD, Principal Investigator — Oncology Department, Ospedale Santa Chiara, Trento; Clorinda Schettino, MD, Study Chair — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No